CLINICAL TRIAL: NCT06927999
Title: An Outpatient, Randomized, Double-Blinded, Placebo-Controlled, Cross-Over Study of the Efficacy of ARS-2 in Patients With Chronic Spontaneous Urticaria
Brief Title: An Outpatient Study of the Efficacy of ARS-2 in Patients With Chronic Spontaneous Urticaria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ARS Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EPI U02
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Urticaria Chronic
MeSH Terms: conditions — Chronic Urticaria | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo solution nasal spray containing no active drug will be administered using the commercial sprayer device.
  Interventions: Drug: Placebo
- 0.5 mg (Active Comparator): 0.5 mg epinephrine per spray
  Interventions: Drug: 0.5 mg epinephrine
- 1 mg (Active Comparator): 1 mg epinephrine per spray
  Interventions: Drug: 1 mg epinephrine

INTERVENTIONS:
Drug: Placebo — Placebo solution nasal spray containing no active drug
  Arms: Placebo
Drug: 0.5 mg epinephrine — 0.5 mg epinephrine per spray
  Arms: 0.5 mg
Drug: 1 mg epinephrine — 1 mg epinephrine per spray
  Arms: 1 mg

SUMMARY:
This is a Phase 2b, outpatient, single-dose, randomized, double blind, placebo-controlled, three period crossover study that will consist of a screening period and three blinded treatment periods. Subjects enrolled will have CSU with a history of moderate to severe acute exacerbations (or flares).

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female between the ages of 18 and 65 years, inclusive.
* Has been clinically diagnosed with CSU and experiences an acute flare of moderate to severe urticaria symptoms (itch and hive severity UAS score ≥ 2) approximately 1-2 times a month or every other month consistently during the past year while on a chronic treatment.
* Has been on a daily chronic treatment for ≥ 6 weeks.
* Is willing to use a smartphone study application to record study assessments and AEs.
* Has body weight more than 15 kilogram (kg).
* Has no medical history of clinically significant hypertension and cardiovascular disease in the last 10 years
* If female, is not pregnant or breastfeeding based on a negative urine pregnancy test at baseline.
* Is able to communicate clearly with the Investigator and staff; able to read, complete questionnaires, and perform study procedures on the smartphone study application.
* Is willing and able to provide written informed consent prior to participating in the study.
* Controlled hypertension without beta blocker confirmed by the Investigator is acceptable.
* At screening, has stable vital signs in the following ranges (after 5 minutes of rest):

  * Systolic blood pressure (SBP) ≥90 and ≤140 milliliters of mercury (mmHg)
  * Diastolic blood pressure (DBP) ≥50 and ≤90 mmHg
  * Heart rate (HR) ≥45 and ≤100 beats per minute (bpm)

Exclusion Criteria:

* Has a history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Has any clinically significant medical condition or PE finding as deemed inappropriate by the Investigator.
* Has abnormal cardiovascular exam at screening including any prior history of myocardial infarction or clinically significant abnormal electrocardiogram (ECG)
* Has had significant traumatic injury or major surgery within 30 days prior to study screening.
* Known hypersensitivity to any compound in the test product, or any other closely related compound (e.g., dihydropyridine-derived molecules).
* Has participated in a clinical trial within 30 days prior to the first dose of study drug.
* Has an immediate family member of the Investigator, or an employee of the study center, with direct involvement in the proposed study, or other studies under the direction of the Investigator or study center or is in a dependent relationship with a study center employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of ARS-2 (0.5 mg or 1 mg) versus placebo on itch and hive | 12 months
  Change in itch and hive scores (Uniform Assessment System) [UAS] as compared to placebo at each timepoint on exacerbation days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Endeavor Health Clinical Trials Center, Glenview, Illinois
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
- Institute of Allergology IFA Charité - Campus Benjamin Franklin | Hindenburgdamm 30, Berlin, Germany